CLINICAL TRIAL: NCT06259773
Title: The Roles of MRI, DYNEELAX and Stress X-ray in First-Line Diagnosis of Cruciate Ligament Injury
Status: Recruiting | Type: Observational
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Yi Ping Wei, Staff doctor, Kaohsiung Veterans General Hospital.
Other Study IDs: 23-CT12-26
Record Dates: First submitted 2024-02-07; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Knee Injuries; Anterior Cruciate Ligament Injuries; Knee Ligament Injury; Knee Arthritis
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: knee stability test (DYNEELAX) — Each knee was tested under a force 120 Newtons in a posterior to anterior direction to create anterior tibial translation at 20 degrees knee flexion. Side-to-side difference of anterior/posterior tibial translation (mm) was measured from radiographs. Measurement of rotation and translation by DYNEELAX was also recorded.

SUMMARY:
Background: Cruciate ligament tears are clinically diagnosed by detection of anterior or posterior tibial translation on physical examination; however, this manual method of assessment is imprecise, subjective, and not reproducible. Recently a new instrument, a stress radiographic device and knee stability test (DYNEELAX), were produced to objectively measure these displacements.

Objective: To assess new diagnostic methods, in the measurement of anterior/posterior tibial translation in cruciate ligament-deficient knee compared to the healthy knee.

Material and method: The MRI, stress radiographic device and knee stability test was applied to cruciate ligament-tear knees that were diagnosed by physical examination as having partial or complete cruciate ligament tears. Each knee was tested under a force 120 Newtons in a posterior to anterior direction to create anterior tibial translation at 20 degrees knee flexion. Side-to-side difference of anterior/posterior tibial translation (mm) was measured from radiographs. Measurement of rotation and translation by DYNEELAX was also recorded.

ELIGIBILITY:
Inclusion Criteria: Patients are diagnoed as ACL/PCL injury or suspect ligament sprain at Kaohsiung veteran general hospital.

Exclusion Criteria: Unable receing MRI exam, any op history of knee or fracture history on the impaired knee.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Over 20 years old, suspected ligament damage caused by knee contusion
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
anterior/posterior tibial translation (mm) | post-op 3 months, 6 months
  by Stress X-ray
patient reported outcome measure | post-op 3 months, 6 months
  Knee Outcome Survey-Activities of Daily Living Score (KOS-ADLS)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ping Wei, Dr., Principal Investigator — Kaohsiung veteran general hospital
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: No